CLINICAL TRIAL: NCT04993859
Title: Impact of Chemotherapy on Urinary Biomarkers and Non-Invasive Urodynamics in Children
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0680.cc; P30CA046934 (NIH); 1K23DK125673-01 (NIH)
Record Dates: First submitted 2021-07-28; First posted 2021-08-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Survivors of Childhood Cancer; Bladder Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Male Cancer Survivors with DVSS Score ≥ 9: Childhood cancer survivors treated with DOX and/or VCR with evidence of BD on DVSS
  Interventions: Diagnostic Test: Non-invasive Urodynamic Test (niUDS); Diagnostic Test: Urinary proteomic screen; Other: Dysfunctional Voiding Symptom Score Survey (DVSS)
- Female Cancer Survivors with DVSS Score ≥ 6: Childhood cancer survivors treated with DOX and/or VCR with evidence of BD on DVSS
  Interventions: Diagnostic Test: Non-invasive Urodynamic Test (niUDS); Diagnostic Test: Urinary proteomic screen; Other: Dysfunctional Voiding Symptom Score Survey (DVSS)
- Male Cancer Survivors with DVSS Score < 9: Childhood cancer survivors treated with DOX and/or VCR without evidence of BD on DVSS
  Interventions: Diagnostic Test: Non-invasive Urodynamic Test (niUDS); Diagnostic Test: Urinary proteomic screen; Other: Dysfunctional Voiding Symptom Score Survey (DVSS)
- Female Cancer Survivors with DVSS Score < 6: Childhood cancer survivors treated with DOX and/or VCR without evidence of BD on DVSS
  Interventions: Diagnostic Test: Non-invasive Urodynamic Test (niUDS); Diagnostic Test: Urinary proteomic screen; Other: Dysfunctional Voiding Symptom Score Survey (DVSS)

INTERVENTIONS:
Diagnostic Test: Non-invasive Urodynamic Test (niUDS) — A noninvasive urodynamics is a simple test used to evaluate urinary flow.
Diagnostic Test: Urinary proteomic screen — Urine proteomics is a powerful platform to identify urinary excreted proteins and peptides in different stages of disease or therapy and to determine their quantity, functions, and interaction.
Other: Dysfunctional Voiding Symptom Score Survey (DVSS) — The Dysfunctional Voiding Symptom Score provides accurate and objective grading of voiding behaviors of children.

SUMMARY:
The over-arching aim of this study is to evaluate the effects of two specific anti-cancer chemotherapies, vincristine and doxorubicin, on bladder function and urine composition.

DETAILED DESCRIPTION:
The over-arching aim of this study is to evaluate the effects of two specific anti-cancer chemotherapies, vincristine and doxorubicin, on bladder function and urine composition. The global hypothesis is that childhood cancer survivors with prior exposure to systemic vincristine (VCR) and/or doxorubicin (DOX) report an increased incidence of bladder dysfunction (BD) symptoms on the Dysfunctional Voiding Symptom Score (DVSS) survey. We expect to observe differences in non-invasive urodynamic (niUDS) testing between childhood cancer survivors with BD symptoms on the DVSS versus those without BD symptoms on DVSS. We also expect to observe statistically significant differences in the urinary levels of known urinary biomarkers of BD (NGF, ATP and BDNF) of patients with evidence of BD compared to those without BD on the DVSS. We also expect to observe rational differences in the urinary proteome of patients between those with and without BD.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-13 years old
* A history of cancer
* Treatment with a chemotherapy regimen including VCR and/or DOX
* Completion of chemotherapy at least one year prior to study enrollment and survey completion.

Exclusion Criteria:

* Patients with a:
* Primary pelvic tumor
* Pelvic irradiation
* Pre-existing bladder/bowel dysfunction
* Spinal defects
* Neurologic disorder
* Neuro-oncologic tumor or brain metastasis
* Cyclophosphamide or ifosfamide therapy

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Study groups and sub-groups will be assigned by gender
Study Population: Childhood cancer survivors that have been treated with a chemotherapy regimen including VCR and/or DOX, completion of chemotherapy at least one year prior to study enrollment and survey completion.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of non-normal niUDS patterns between groups | Immediately after niUDS done at the first visit
  a. Patterns will be scored by blinded reviewers b. Will calculate an Inter-rater Kappa correlation co-efficient i. Utilize consensus review for discrepancies between reviewers and between the patient's 1st/2nd niUDS for the final assignment ii. Will calculate an intra-test reliability (compare correlation between 1st and 2nd patter) c. Chi-square test to compare proportions of non-normal vs. normal pattern type i. Group 1a vs. 2a ii. Group 1b vs. 2b d. Sample Size Calculation: Based on published data of niUDS patterns in children with normal bladder function, we expect 15% of those children in Group 2 to have non-normal niUDS patterns. We hypothesize that 40% of children in Group 1 to have non-normal niUDS patterns. 38 subjects in each gender sub-group provide 80% power to detect this 25% difference with an one-sided chi-square test with an alpha of 0.05.
Proportion of Elevated Post-Void Residual (PVR) between groups | 13 months
  a. Will use an "average PVR" between the 1st/2nd niUDS for the analysis b. Chi-square test to compare proportions of elevated PVR i. Group 1a vs. 2a ii. Group 1b vs. 2b c. Sample Size Calculation: Based on published data of PVR in children with normal bladder function, we expect 1.5% of those children in Group 2 to have elevated PVR. We hypothesize that 25% of children in Group 1 to have an elevated PVR. 21 subjects in each gender sub-group provide 80% power to detect this 23.5% difference with an one-sided chi-square test with an alpha of 0.05.
Compare Peak Flow Rates (Qmax) between groups | 13 momths
  a. Will use the average of the two Qmax between the 1st/2nd flow rate for the analysis b. Two group t-test for comparing continuous variables (Qmax) i. Group 1a vs. 2a ii. Group 1b vs. 2b c. Sample Size Calculation: 38 subjects in Group 1a and 2a provide 80% power to detect an effect size of 0.7 (mean difference divided by the common standard deviation) using a 2-sided two-group test with an alpha of 0.05. if the outcome is not normally distributed, transformation will be carried out so the distribution will be approximately normal. This power calculation also applies to the comparison between Group 1b vs 2b
Compare Average Flow Rates (Qavg) for age/gender | 13 months
  a. Will use the average of the two Qavg between the 1st/2nd flow rate for the analysis b. Two group ttest for comparing continuous variables (Qavg) i. Group 1a vs. 2a ii. Group 1b vs. 2b c. See the power calculation in 3c.
Compare Urinary Biomarker Levels between groups | 13 months
  1. Compare urinary biomarker levels between groups i. ATP, BDNF, NGF ii. Two-group t-test for comparing continuous variables
  1. Group 1 vs. 2
  2. Sub-analysis
     1. Group 1a vs. 2a
     2. Group 1b vs. 2b The sample size calculation in 1d can apply to each biomarker. Based on published data in other populations with BD, for NGF, ATP and BDNF, we hypothesize to detect a difference of these urinary biomarkers 2x higher in Group 2 (Elevated DVSS scores) vs. Group 1 (Normal DVSS scores).
  A mixed effects model will be used to estimate and compare a biomarker expression between the two groups by incorporating the individual measurements on each subject into the model, where gender and group assignment will be the predictor. Interaction term between group and gender will be considered to study the effect modification by gender on a biomarker if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Cost, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient Data will be shared after written request to study PI and after approval by local IRB and study committee
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after publication, for a total of 5 years
Access Criteria: Written proposal with IRB approval